CLINICAL TRIAL: NCT03864809
Title: • Sleep Disturbance Among Patients With Psoriasis and Atopy and Comparison Between Them
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amani Mahmoud Abdelmohsen, Principal Investigator, Assiut University
Other Study IDs: SL disturb in psoriasis atopy
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- psoriasis patients: sleep disturbance
  Interventions: Behavioral: sleep disturbance
- atopic dermatites patients: sleep disturbance
  Interventions: Behavioral: sleep disturbance
- control: sleep disturbance
  Interventions: Behavioral: sleep disturbance

INTERVENTIONS:
Behavioral: sleep disturbance — we observe sleep disturbance among patients with psoriasis and atopic dermatitis and control group

SUMMARY:
Comparison between sleep disturbance in atopy and psoriasis and control

DETAILED DESCRIPTION:
Sleep is essential for daytime functioning and health and important for both psychological and physiological wellbeing . A growing body of research indicates that chronic sleep disturbance is associated with impaired quality of life (QoL) and a risk factor for poorer health, for example depression cardiovascular disease, hypertension 1 and diabetes.

insomnia, the most common sleep disorder, is a clinical condition defined as difficulties falling asleep and/or maintaining sleep and/or poor sleep quality despite adequate opportunity for sleep resulting in significant daytime impairment.

The development of insomnia in healthy populations has a bi-directional relationship with psychological factors such as anxiety, depressive symptoms and stress, and may in clinical populations also be associated with physical symptoms, such as pain. the physical symptoms in psoriasis, such as itch, one would expect a higher prevalence of sleep disturbance in this patient group. On the other hand Sleep disturbance is common also in patients with atopic dermatitis (AD). Patients with AD often have sleep disturbances due to pruritus.

ELIGIBILITY:
Inclusion Criteria:

- patients with Psoriasis and Patients with A topic dermatitis

Exclusion Criteria:

* All patient have another dermatological disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study involves the use of seven questionnaires to be given to subjects with psoriasis and a topic dermatites
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
severity of the psooriasis (Psoriasis Area and Severity Index) | 1 hour
  calculation of the severity through questionaire , 0 = None
  1. = Slight
  2. = Moderate
  3. = Severe
  4. = Very severe

SECONDARY OUTCOMES:
2.HRQoL (Dermatology Life Quality Index); | 1 hour
  The aim of this questionnaire is to measure how much your skin problem has affected your life OVER THE LAST WEEK The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
.insomnia severity [Insomnia Severity Index (ISI)]; | 1 hour
  The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score. When you have your total score
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
sleep quality [Pittsburgh Sleep Quality Index (PSQI)]; | 1 hour
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
  A total score of "5" or greater is indicative of poor sleep quality. If you scored "5" or more it is suggested that you discuss your sleep habits with a healthcare provider
stress (Perceived Stress Scale); | 1 hour
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful.
  0 = Never 1 = Almost Never 2 = Sometimes 3 = Fairly Often 4 = Very Often
itch (Itch Severity Scale); | 1 hour
  The ISS consists of seven questions that measure the severity of itch and the extent to which QoL is affected. The total score ranges from zero to 21
and depressive symptoms (Beck Depression Inventory | 1 hour
  This depression inventory can be self-scored 1-10____________________These ups and downs are considered normal 11-16___________________ Mild mood disturbance 17-20___________________Borderline clinical depression 21-30___________________Moderate depression 31-40___________________Severe depression over 40__________________Extreme depression
severity of a topic dermatitis | 1 hour
  The eczema area and severity index (EASI) Mild eczema score < 25 Moderate eczema score >25 <50 Severe eczema score >50

CONTACTS AND LOCATIONS:
Overall Officials: radwa bakr, lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Jensen P, Zachariae C, Skov L, Zachariae R. Sleep disturbance in psoriasis: a case-controlled study. Br J Dermatol. 2018 Dec;179(6):1376-1384. doi: 10.1111/bjd.16702. Epub 2018 Aug 23. PMID 29704428